CLINICAL TRIAL: NCT03763448
Title: Effects of Infrapatellar Fat Pad Preservation Versus Resection on Clinical Outcomes After Total Knee Arthroplasty in Patients With Knee Osteoarthritis - A Multicenter Randomized Controlled Clinical Trial
Brief Title: Infrapatellar Fat Pad Preservation Versus Resection on Clinical Outcomes After Total Knee Arthroplasty(IPAKA)
Acronym: IPAKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Peking University People's Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); First Affiliated Hospital of Jinan University (Other); Anhui Provincial Hospital (Other Government); Tianjin Hospital (Other); Youjiang Medical College for Nationalities (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Ding Changhai, Director,Clinical Research Center, Zhujiang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-GJGBK-001
Record Dates: First submitted 2018-10-19; First posted 2018-12-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis; Arthropathy of Knee
Keywords: Infrapatellar Fat Pad; Knee Osteoarthritis; Total Knee Arthroplasty; Randomized Clinical Trial
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participants, outcome assessors, data analysts and chief investigators are masked during the study procedure.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infrapatellar Fat Pad Preservation (Experimental): The IPFP retention of more than 80% in actual operation shall be regarded as IPFP retention.
  Interventions: Procedure: Infrapatellar Fat Pad preservation
- Infrapatellar Fat Pad Resection (Active Comparator): In the clinical practice, more than 80% of IPFP volume is commonly resected by surgeons during total knee arthroplasty. The investigators hereby define resection of more than 80% IPFP volume as IPFP excision.
  Interventions: Procedure: Infrapatellar Fat Pad resection

INTERVENTIONS:
Procedure: Infrapatellar Fat Pad preservation — In the IPFP preservation group, IPFP (more than 80%) will be preserved by retracting out of the operative field.
  Other Names: Infrapatellar fat pad retention
  Arms: Infrapatellar Fat Pad Preservation
Procedure: Infrapatellar Fat Pad resection — In the IPFP resection group, more than 80% IPFP will be resected during the total knee arthroplasty.
  Arms: Infrapatellar Fat Pad Resection

SUMMARY:
This study aims to compare the postoperative clinical outcomes of Infrapatellar Fat Pad (IPFP) preservation versus resection after total knee arthroplasty (TKA) in patients with knee osteoarthritis. Participants will be identified as normal IPFP or abnormal IPFP based on MRI findings before randomization. The primary outcome is the change from baseline to 12 months in the mean score on five Knee Injury and Osteoarthritis Outcome Score (KOOS) subscales (KOOS5), covering pain, symptoms, activities of daily life, sport & recreation, knee-related quality of life, with scores ranging from 0 (worst) to 100 (best). The secondary endpoints will be included: KOOS subscales, Knee Society Score (KSS), 100 mm Visual Analogue Scale (VAS) Pain, timed up-and-go test, depression, patellar tendon shortening, 100 mm VAS self-reported efficacy of reduced pain and increased quality of life. Adverse events will be recorded. Primary and secondary outcomes will be evaluated or reported blindly at baseline and at postoperative 3 months, 6 months, and 1 year. Intention-to-treat analyses will be used.

DETAILED DESCRIPTION:
Knee Osteoarthritis (KOA) is a common chronic disease, which often leads to joint pain and limited function in the elderly, and thus affects participants' quality of life. Total knee arthroplasty (TKA) has been developed as a mature surgical procedure to relieve end-stage osteoarthritic joint pain and improve limb function. Although more than 80% of the patients reported in the literature are satisfied with the postoperative efficacy of TKA, there are still a large number of patients whose daily life is affected by persistent knee pain and limited function after the operation of the affected limb.

The IPFP is a fat mass located behind the patellar ligament, between the lower part of the patella and the tibial tubercle. The function of IPFP is controversial at present. It is reported that IPFP can provide blood supply for anterior cruciate ligament, patella and patellar ligament through the arterial network of the knee joint. In addition, it can fill the joint gap to lubricate the surface of the joint, reduce friction and absorb impulse so as to play a physiological protective role. On the contrary, studies have pointed out that abnormal IPFP could produce various pro-inflammatory cytokines such as interleukin (IL)-1β, tumour necrosis factor (TNF)-α, IL-6 and IL-8, as well as adipokines such as leptin and resistin, and thus might play a detrimental role in knee OA. Traditionally, the IPFP has been removed in order to improve surgical exposure and to prevent interposition during baseplate implantation. Despite the significant evolution of TKA technology which no longer requires the resection of IPFP for better surgical access, IPFP is still partially or totally resected in around 88% of TKAs.

The investigators' previous population-based cohort study revealed that IPFP maximal area and volume were associated with reduced knee pain, decreased loss of cartilage volume and reduced risks of cartilage defect progression, indicating a beneficial effect of IPFP size. On the other hand, the investigators' further investigation demonstrated that IPFP signal intensity alteration was negatively associated with maximum area of IPFP, and moreover, associated with increased knee cartilage defects, subchondral bone marrow lesion (BML) and knee pain, suggesting IPFP with abnormal quality may play a detrimental role in knee OA. Based on these findings, the investigators proposed that IPFP with normal quality should be preserved or not damaged during TKA, while IPFP with abnormal quality should be resected. This multicentre randomised controlled trial is designed to test the investigators' hypotheses: in patients with normal IPFP quality, preservation of IPFP during TKA procedure will reduce postoperative knee symptoms and improve joint function, comparing with IPFP resection during TKA procedures; in patients with abnormal IPFP quality, resection of IPFP during TKA procedure will reduce postoperative knee symptoms and improve joint function, comparing with IPFP preservation during TKA procedures. The results would provide evidence-based recommendations on clinical practice to improve OA patients' postoperative outcomes.

Three hundred and sixty eligible participants will be recruited and identified as having normal IPFP quality (signal intensity alteration score ≤ 1) or abnormal IPFP quality (signal intensity alteration score ≥ 2). Participants in each site will be randomly allocated to IPFP resection group or preservation group using computer-generated block randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with knee osteoarthritis by X-ray plain film (Kellgren-Lawrence score of ≥ 2)
* The need for TKA was confirmed after evaluation by the orthopedic surgeon
* One week before surgery, knee pain 100mm pain visual analogue scale score was greater than 20mm
* Understanding of the study requirements and willing to participate in this study

Exclusion Criteria:

* Rheumatoid arthritis,psoriatic arthritis,lupus,malignant tumor
* Requiring contralateral TKA within one year
* The visual analogue score of 100mm of knee pain before operation was less than 20mm
* Having a possible or planned pregnancy
* With poor compliance
* Suffering from somatic disease, psychiatric or cognitive disorders, neurological disorders that will compromise the safety, compliance, consent, participation, follow-up and the interpretation of the results
* Severe knee valgus
* Contraindications with TKA or MRI

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
The mean score on five Knee Injury and Osteoarthritis Outcome Score(KOOS) subscales | From pre-operation to 12 months after operation
  The primary outcome was the change from baseline to 12 months in the mean score on five Knee Injury and Osteoarthritis Outcome Score (KOOS) subscales, covering pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life (KOOS5), with scores ranging from 0 (worst) to 100 (best). The KOOS, a valid, reliable and responsive self-reported questionnaire applied to evaluate the short and long-term patient-relevant outcomes following TKA, consists of five subscales with a total of 42 items: pain (9 items), symptoms (7 items), function in ADL (17 items), sport and recreation function (5 items) and knee-related quality of life (4 items).

SECONDARY OUTCOMES:
Five individual subscales of Knee Injury and Osteoarthritis Outcome Score (KOOS) | From pre-operation to 12 months after operation
  KOOS subscales including pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. Scores are transformed to a 0-100 scale, with 0 representing worst health and 100 representing best health.
Knee Society Score(KSS) | From pre-operation to 12 months after operation
  KSS is a rating system that consists of two scores: joint score and functional score. Both scores range from 0 (worst health or functioning) to 100 (best health or functioning).
Self-reported efficacy of reduced pain and increased quality of life | From pre-operation to 12 months after operation
  Using a 100mm VAS with terminal descriptors of "very unsure" and "very sure"
Insall - Salvati Ratio (ISR) | From pre-operation to 12 months after operation
  It is used to assess changes in the length of the patellar tendon at baseline and month 12. Lateral radiographs with the knee in about 30 degree of flexion will be taken by well experienced X-ray technicians using standardized radiographic techniques. The numerator of the ISR-the length of the patellar tendon-was determined by measuring the distance from inferior aspect of the patella to the superior aspect of the tibial tubercle. The longest dimension of the patella on the lateral radiograph will be obtained as denominator of the ISR.
Timed Up and Go test | From pre-operation to 12 months after operation
  It is a simple test used to assess a person's mobility. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Visual Analogue Scale (VAS) Pain | From pre-operation to 12 months after operation
  Pain intensity measured on a 100 mm VAS with terminal descriptors of "no pain" and "worst pain possible" in the following situations: at rest, after 30-min of walking, and on most days of the last month.

CONTACTS AND LOCATIONS:
Overall Officials: Changhai Ding, MD, Principal Investigator — Clinical Research Center of Zhujiang Hospital,Southern Medical University; Jianhao Lin, MD, Principal Investigator — Peking University People's Hospital; Xisheng Weng, MD, Principal Investigator — Peking Union Medical College Hospital; Guanghua Lei, MD, Principal Investigator — Xiangya Hospital of Central South University; Zongsheng Yin, MD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University; Zhengang Zha, MD, Principal Investigator — First Affiliated Hospital of Jinan University; Jing Tian, MD, Principal Investigator — Zhujiang Hospital; Xifu Shang, MD, Principal Investigator — Anhui Provincial Hospital; Yujin Tang, MD, Principal Investigator — Youjiang Medical College for Nationalities; Jun Liu, MD, Principal Investigator — Tianjin Hospital
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhu Z, Han W, Lu M, Lin J, Yin Z, Shang X, Weng X, Zha Z, Tian J, Lei G, Hunter DJ, Ding C. Effects of infrapatellar fat pad preservation versus resection on clinical outcomes after total knee arthroplasty in patients with knee osteoarthritis (IPAKA): study protocol for a multicentre, randomised, controlled clinical trial. BMJ Open. 2020 Oct 23;10(10):e043088. doi: 10.1136/bmjopen-2020-043088. PMID 33099502